CLINICAL TRIAL: NCT00225602
Title: Quasi-Experimental Trial of the Effect of Assertive Community Treatment Among Those With Severe Mental Disorder
Brief Title: Assertive Community Treatment in Copenhagen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Copenhagen Hospital Corporation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBH363004; Cph Hospital Corporation; Østdansk Forskningsforum
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2005-09-26 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; Assertive community treatment
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Community Mental Health Services; Therapeutics; Community Mental Health Centers

INTERVENTIONS:
Behavioral: Assertive Community Treatment
Behavioral: Treatment in Community Mental Health Center

SUMMARY:
The aim of the study is to evaluate the effect of assertive community treatment in Copenhagen in two regions compared with two regions where this treatment was not implemented. The effect on user satisfaction, use of bed days, social network, global assessment of functioning, substance misuse will be evaluated.

DETAILED DESCRIPTION:
In area where assertive community treatment was implemented 100 patients had filled in a form regarding their social situation. They were interviewed after one year and asked about user satisfaction and followed up in Danish registers. Register information was extracted concerning vital status, cause of death, use of psychiatric services and criminal record. The same procedure was carried out for a comparison group, carefully matched, from other regions in Copenhagen, where assertive community treatment was not implemented.

ELIGIBILITY:
Inclusion Criteria:

* User of bed days exceeded 40 days last two years; or
* 4+ admissions during last two years; or
* A second diagnosis of substance misuse; or
* Non compliance with medication or outpatient visits in usual settings; or
* Being unable to use other existing services

Exclusion Criteria:

* Forensic patient with a sentence to stay in hospital

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Adherence to treatment

SECONDARY OUTCOMES:
Experience of violation of personal integrity and privacy in relation to treatment
User satisfaction
Quality of Life
Substance misuse
Social network
Affiliation to labor market
Independent living
Crime
Suicidal behaviour
Use of psychiatric services

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Ph.D, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen, Denmark